CLINICAL TRIAL: NCT01508559
Title: Neurocognitive Function in a Central London Cohort of HIV Infected and Uninfected Men Who Have Sex With Men
Brief Title: Men Who Have Sex With Men (MSM) Neurocog 1&2 Study
Acronym: MSM Neurocog
Status: Completed | Type: Observational
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Other Study IDs: MSM Neurocog
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: HIV Related Neurocognitive Impairment
Keywords: HIV; Neurocognitive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV infected: HIV infected MSM 18-50 years old
- HIV uninfected: HIV uninfected MSM 18-50 years old

SUMMARY:
The treatment of HIV and the tests performed for HIV care have changed over the last 20 years but improvement of management of HIV-infected subjects is still warranted. The investigators would like to collect and analyse clinical information obtained from subjects who are between 18 and 50 years of age. The investigators will look at routine clinic information such as blood pressure, recent blood test results and clinical history. The investigators will then assess cognitive (brain) function by talking and/or written tests. These tests will include tests for memory, depression and anxiety.

All of those who are identified as having problems with their brain function in this way will be offered onward referral for further assessment as appropriate. Those taking part will be offered a follow up visit at 24-48 weeks after the first assessment to see if there are any changes. This will allow us to understand how brain problems develop, get worse, or get better over time. No genetic research will be done. Depression is a mental health condition that can be characterized by negative feelings, a generally low mood, or problems with eating and sleeping normally. Anxiety is also a mental health condition where a person can feel general anxiousness or fear of specific situations, or, in more serious cases, can have panic attacks. Impaired brain function is a condition of the nervous system or brain where the brain does not function as well as it normally should, and can include symptoms such as forgetfulness, doing everyday tasks more slowly or becoming disorientated to the time of day or the place one is in.

For this study, the investigators will also collect data from medical records, including (and if known)social and educational-related data, HIV infection-related data (e.g. date of diagnosis, blood test results), relevant medical history (e.g. previous psychiatric conditions) and medication used (e.g. date started, the drugs used).

The information the investigators will get from this study will be used to inform healthcare providers (doctor, nurse, health advisor, psychologist) on whether it is necessary to routinely assess HIV infected patients for the presence of anxiety/depression and impaired brain function. The investigators will also get information on whether the treatments used for HIV infection make a difference to how commonly these conditions occur in patients.

DETAILED DESCRIPTION:
The aim of this project is to examine neurocognitive functioning in HIV infected men who have sex with men (MSMs). We have limited our study to this group in order to better study other shared risk factors (hepatitis coinfection, recreational drug use). Given ongoing work in an older cohort our aim is to study neurocognitive impairment in younger subjects (18-49 years). There are two parts to this study. The first is a cross sectional pilot (MSM Neurocog-1) looking at neurocognitive function in HIV infected and HIV uninfected MSMs. The second plan is for a prospective 48 week cohort study 24-48 week study (MSM Neurocog-2) following neurocognitive function in HIV infected subjects and a group of HIV uninfected controls over time.

The shift in HIV care to that of a chronic, manageable condition has transferred focus to long-term morbidities and drug toxicities. One such area in which there is renewed interest is the prevalence and relevance of neurocognitive impairment, as well as the significance of compartmentalised virus in the CSF as compared to blood. Controlled, comparative data are lacking - many of the cross-sectional studies to date have not controlled for important confounders such as recreational and injecting drug use, current or prior co-infections or co-morbidities. Where this has happened, researchers generally use general population controls that may differ markedly from HIV-infected individuals in terms of lifestyle and demographic factors. In addition the paucity of longitudinal data means it is unclear whether an individual with normal neurocognitive function pre-ART will develop impairment later or if subjects with evidence of impairment can expect improvement or normalisation over time; these issues are highly important for clinical management and patient counselling. There is no consensus on which surrogate markers, if any, are important in terms of diagnosing, monitoring and/or predicting neurocognitive impairment. Studies measuring correlation between neurocognitive performance and neuronal markers of inflammation have been conflicting.

ELIGIBILITY:
Inclusion Criteria:

All subjects

* 18-49 years inclusive
* Identifying as MSM
* Willing and able to provide written informed consent
* Able to complete screening tools.
* Fluent in spoken and written English
* Patients who have given written and dated informed consent to participate in this study and to use the data.
* Patients co-infected with chronic hepatitis B/C (diagnosed serologically at least 6 months prior to study to exclude seroconversion/recent infection) and/or currently using recreational substances including alcohol will be included in this study ("real world" data)

HIV-infected subjects • Known HIV of at least 6 months duration (in order to exclude symptoms associated with primary HIV infection)

HIV-uninfected controls

* HIV-negative by rapid point of care test (POCT) or standard laboratory testing
* No unprotected anal intercourse (UPAI) in last 3 months

Exclusion Criteria:

All subjects

* HIV or hepatitis B/C infection thought to have occurred in the last 6 months
* Current/active central nervous system (CNS) opportunistic infections or CNS malignancies.
* Previous cerebrovascular accidents (CVA/stroke) or history of transient ischemic attacks (TIAs).
* Neuromuscular disease that will limit ability to perform the screening tests.
* Patients receiving current therapy with ribavirin or interferon for hepatitis co-infection or expected to start such therapy in the coming 12 months
* Current medical or psychiatric/psychological condition deemed significant by the investigator o (e.g. psychosis, bipolar disorder, dementia, eating disorders, severe head injury (loss of consciousness for at least an hour), current CNS opportunistic infection)

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: HIV infected and uninfected MSM 18-50 years old
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Neurocognitive screening score | 0-6 months
  To describe the prevalence of a positive screening for neurocognitive impairment (NCI) HIV infected and uninfected men who have sex with men (MSM) population using the Basic Neurocognitive Score (BNCS) and International HIV Dementia Score (IHDS) as validated screening tools
Change in neurocognitive function | 0-6 months
  To follow neurocognitive function over time in a cohort of HIV infected and uninfected MSMs

SECONDARY OUTCOMES:
Demographics | 0-6 months
  To explore possible correlations between baseline demographics and disease characteristics and prevalence of positive screens for anxiety and/or depressive symptoms and NCI
Biomarkers | 0-6 months
  To look for possible markers of NCI on MRI scanning or on serological/CSF analysis

CONTACTS AND LOCATIONS:
Overall Officials: Brian Gazzard, Prof, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- SSAT Clinical Trials Unit, London, United Kingdom